CLINICAL TRIAL: NCT00696501
Title: Direct Stimulation Of Spinal Nerve Roots To Determine Sensory And Motor Innervation Patterns
Status: Terminated | Type: Observational
Why Stopped: One of the investigators left the Institution
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-039
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Spine Surgery; Neuromuscular Mapping; Neurodiagnostics
Keywords: Neuromuscular mapping; Spinal surgery; Neurodiagnostics; Segmental root innervation; Dermatomal innervation; Myotomal innervation; Nerve roots; Sensory; Signs and Symptoms
MeSH Terms: conditions — Signs and Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect data while monitoring muscles and nerves during spine surgery. The data being collected and analyzed will be used to learn more about how the body's nerves and muscles are distributed and develop a map of human muscle innervation patterns.

DETAILED DESCRIPTION:
In this large scale study it is proposed to examine root-to-muscle innervation directly, using the standard Intra-Operative Monitoring procedures during scheduled cervical and lumbar spinal surgeries. The study would directly map muscle and sensory distributions of nerve root innervations with no additional risk to patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing either cervical or lumbar cord procedures at Lahey Clinic and during which the surgeon has requested intra-operative neurophysiologic monitoring.
* Surgery performed by a neurosurgeon
* Participant must be ≥ 18 years of age or ≤ 85 years of age
* Participant, or legally authorized representative, has been informed of the nature of the study and has provided written informed consent, approved by the Lahey Clinic IRB

Exclusion Criteria:

Past medical history significant for any of the following:

* Peripheral Neuropathy
* Patients with Diabetes Mellitus
* Neuromuscular disease that would interfere with intra-operative recordings
* The Investigator determines that the patient should not be included in the study for reason(s) not already specified

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All neurosurgical patients will be screened for potential eligibility from the Neurosurgery Department's Clinical and operative schedules.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2006-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Build a database of spinal nerve root innervation utilizing direct nerve root stimulation | Data collected during surgery and a 30 day post-op visit

SECONDARY OUTCOMES:
Compare clinical symptoms of the patient to the direct muscle activation via spinal nerve root stimulation | Data collected during surgery and a 30 day post-op visit

CONTACTS AND LOCATIONS:
Overall Officials: Subu N. Magge, M.D., Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Neurosurgery Department, Lahey Clinic, Inc., Burlington, Massachusetts, United States

REFERENCES:
- [Background] Dykes RW, Terzis JK. Spinal nerve distributions in the upper limb: the organization of the dermatome and afferent myotome. Philos Trans R Soc Lond B Biol Sci. 1981 Aug 12;293(1070):509-54. doi: 10.1098/rstb.1981.0083. PMID 6115429
- [Background] Tsao BE, Levin KH, Bodner RA. Comparison of surgical and electrodiagnostic findings in single root lumbosacral radiculopathies. Muscle Nerve. 2003 Jan;27(1):60-4. doi: 10.1002/mus.10291. PMID 12508296
- [Background] Levin KH, Maggiano HJ, Wilbourn AJ. Cervical radiculopathies: comparison of surgical and EMG localization of single-root lesions. Neurology. 1996 Apr;46(4):1022-5. doi: 10.1212/wnl.46.4.1022. PMID 8780083
- [Background] Moller AR. Intraoperative neurophysiologic monitoring. Am J Otol. 1995 Jan;16(1):115-7. No abstract available. PMID 8579167
- [Background] Bose B, Sestokas AK, Schwartz DM. Neurophysiological monitoring of spinal cord function during instrumented anterior cervical fusion. Spine J. 2004 Mar-Apr;4(2):202-7. doi: 10.1016/j.spinee.2003.06.001. PMID 15016399
- [Background] MacDonald DB. Safety of intraoperative transcranial electrical stimulation motor evoked potential monitoring. J Clin Neurophysiol. 2002 Oct;19(5):416-29. doi: 10.1097/00004691-200210000-00005. PMID 12477987
- [Background] Deletis, V. (2002), Intraoperative Neurophysiology and Methodologies Used to Monitor the Functional Integrity of the Motor System
- [Background] Chiappa, K.H. (1997) Evoked Potentials in Clinical Medicine